CLINICAL TRIAL: NCT06429319
Title: An Open-label Multicenter Postmarketing Extension Study of Efficacy and Safety of Intra-articular HBISA Endoprosthesis of Synovial Fluid NOLTREX™ in Knee Osteoarthritis
Brief Title: Intra-articular Polyacrylamide Hydrogel in Gonarthrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Centre BIOFORM (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IA/PAAG-SI/OA/2020
Record Dates: First submitted 2020-08-14; First posted 2024-05-24 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis
Keywords: intra-articular; polyacrylamide hydrogel; PAAG; HBISA (Hydrous biopolymer with silver ions "Argiform"); NOLTREX
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: This was an open-label extension (OLE) of the IA/PAAG-SI/OA/2019 study designed to evaluate the long-term safety and efficacy of MD NOLTREX™ in patients with knee osteoarthritis (OA). The study was expected to enroll 72 patients who had completed the parent study. Actually 67 patients rolled over into the OLE, 2 of them were classified as screen failures and 65 were enrolled into the trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medical Device: HBISA (polyacrylamide hydrogel) synovial fluid endoprosthesis NOLTREX™ (Other): Sixty-five (65) patients were included in the study and divided into three groups based on the number of NOLTREX™ courses received:
  * Group A consisted of 5 patients who received 2 NOLTREX™ courses, the first course in the IA/PAAG-SI/OA/2019 study and the second one at Visits 1/2 of OLE (IA/PAAG-SI/OA/2020) study.
  * Group B comprised 43 patients who received 2 NOLTREX™ courses, the first course in the IA/PAAG-SI/OA/2019 study and the second one at Visits 3/4 of OLE.
  * Group C consisted of 17 patients who had received only 1 NOLTREX™ course in the parent study.
  Interventions: Device: Hydrous biopolymer with silver ions "Argiform" (HBISA) endoprosthesis of synovial fluid NOLTREX™

INTERVENTIONS:
Device: Hydrous biopolymer with silver ions "Argiform" (HBISA) endoprosthesis of synovial fluid NOLTREX™ — If clinically indicated patients received a repeat course of NOLTREX™ (one or two weekly intra-articular injections of 4.0 NOLTREX™ at the investigator's discretion depending on the stage of OA and clinical response to treatment).
  Other Names: Polyacrylamide hydrogel with silver ions

SUMMARY:
The OLE was aimed to assess long-term safety and efficacy of one and two courses of IA HBISA in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
HBISA (polyacrylamide hydrogel) endoprosthesis of synovial fluid NOLTREX™ is intended for the symptomatic treatment of adult patients with osteoarthritis (OA) reducing pain and improving mobility.

The aim of the 6-month OLE was to evaluate the long-term safety and efficacy of one and two courses of IA Polyacrylamide hydrogel with silver ions in patients with knee osteoarthritis who had received at least one IA injection of NOLTREX™ and completed the visit 5 in the IA/PAAG-SI/OA/2019 study.

In OLE patients who had received a course of treatment (one or two weekly intra-articular injections of 4.0 NOLTREX™ depending on the stage of OA and the clinical response to treatment) in the parent study might receive a single repeat course of NOLTREX™ at the visits 1/2 or 3/4 when clinically indicated. The WOMAC was the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 50 years of age;
* Provision of signed informed consent form;
* Patients met ACR classification criteria for knee osteoarthritis (pain in the knee and at least three of the following: age >50 years, stiffness <30 min, crepitus, bony tenderness, bony enlargement and no palpable warmth);
* OA grades 2 and 3 on the Kellgren-Lawrence scale with the predominant involvement of the medial tibiofemoral region of the knee joint;
* Patients from the NOLTREX™ group of the parent study (IA/PAAG-SI/OA/2019) who completed all (5) study visits

Exclusion Criteria:

1. Pregnancy and breastfeeding;
2. History of trauma or surgery on the target knee joint;
3. Instability of the target knee joint;
4. Microcrystalline arthropathies (according to the history and taking into account clinical manifestations);
5. History of systemic inflammatory diseases (rheumatoid arthritis, systemic lupus erythematosus, etc.);
6. Seronegative spondyloarthritis and reactive arthritis;
7. Increased rheumatoid factor;
8. Increased uric acid > 360 µmol/l;
9. Intra-articular injection into the target knee joint:

   * hyaluronates - within 12 months prior to patient enrollment in the study;
   * other synovial fluid endoprostheses (except for NOLTREX™ in the IA/PAAG- SI/OA/2019 study) within 24 months;
   * glucocorticoids - within 1 month before enrollment in the study;
   * NSAIDs - intra-articular injection at any time in the history.
10. Systemic pain medications (NSAIDs, opioid analgesics) within 1 week prior to Visit 0;
11. Effusion in the target joint;
12. The presence of inflammation or infection in the target joint, synovitis;
13. The need for continuous use of glucocorticoids in any dosage form;
14. Use of paracetamol within 48 hours prior to Visit 0;
15. A positive blood test result for one or more of the following infections: HIV, hepatitis B and C, syphilis;
16. Severe liver disease, defined as an increase in one of the following: ALT, AST, alkaline phosphatase, total bilirubin, GGT more than 3 times the upper limit of normal;
17. Kidney disease with a glomerular filtration rate as assessed by the Cockcraft-Gault formula less than 60 mL/min/1.73 m2 (stages III-V chronic kidney disease [CKD]);
18. Clinical manifest coxarthrosis;
19. Severe decompensated chronic or acute diseases and other conditions or other causes that, in the investigator's opinion, may prevent the patient from participating in the study or affect the study results ;
20. Participation in any other clinical trial except that IA/PAAG-SI/OA/2019 within 90 days prior to enrollment in the OLE.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2021-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir V Popov, DSc, Principal Investigator — Non-budgetary HCF "Railway clinical hospital n.a. Semashko N.A. at Lublino, OJSC "Russian Railways"
Locations (4):
- Russia (4):
  - Non-budgetary healthcare facility "Railway clinical hospital n.a. Semashko N.A. at Lublino, OJSC "Russian Railways", Moscow
  - "Clinical Diagnostic Center "Ultramed", LLC, Omsk
  - Private Healthcare Facilty "Clinical hospital "RZHD-Medicina" of the city Saint-Petersburg, Saint Petersburg
  - State budgetary healthcare facility of Yaroslavl Region "Clinical hospital №3", Yaroslavl

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Group A consisted of 5 patients who received 2 NOLTREX™ courses, the first course in the parent (IA/PAAG-SI/OA/2019) study and the second one at Visits 1/2 of the OLE (IA/PAAG-SI/OA/2020) study.
- Group B: Group B comprised 43 patients who received 2 NOLTREX™ courses, the first course in the parent (IA/PAAG-SI/OA/2019) study and the second one at Visits 3/4 of OLE.
- Group C: Group C consisted of 17 patients who had received only 1 NOLTREX™ course in the parent study.
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 5 | 43 | 17
Completed | 5 | 43 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were described by group in the safety population (SP). The safety population was the same as the ITT population and included all randomised patients.
Groups:
- Group A: Group A consisted of 5 patients who received 2 NOLTREX™ courses, the first course in the IA/PAAG-SI/OA/2019 study and the second one at Visits 1/2 of OLE (IA/PAAG-SI/OA/2020) study.
- Group B: Group B comprised 43 patients who received 2 NOLTREX™ courses, the first course in the IA/PAAG-SI/OA/2019 study and the second one at Visits 3/4 of OLE.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 5 | 43 | 17 | 65
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 71.60 (11.15) | 63.53 (5.93) | 61.88 (7.27) | 63.72 (7.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 37 | 11 | 53
  Male | 0 | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 43 | 17 | 65
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.28 (2.32) | 28.97 (3.15) | 27.18 (1.82) | 28.68 (2.98)
Obesity [Count of Participants; unit: Participants] | 4 | 14 | 1 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in the Total WOMAC Score (WOMAC-T)
Description: Mean change in WOMAC-T from baseline (visit 0 [screening] of OLE and visit 1 (week 1) of the parent study) to visit 3 (week 11) and visit 5 (week 23). Patients were asked to complete the questionnaire during the study visits. The Western Ontario and McMaster Universities Osteoarthritis Index Version 3.1 Visual Analog Scale Format (WOMAC VA 3.1) applies a 100-mm VAS and consists of three subscales: pain (5 questions), stiffness (2 questions), and physical function (17 questions). The scores for each subscale are summed up, with a possible score range of 0-500 for Pain, 0-200 for Stiffness, and 0-1700 for Physical Function. Higher scores represent worse pain, stiffness, and functional limitations. A sum of the scores for all three subscales gives a total WOMAC score (0-2400), where 0 represents the best and 2400 the worst possible health status. The higher the score, the poorer the function. Therefore, an improvement was achieved by reducing the overall score.
Time Frame: baseline (OLE visit 0 and visit 1 study 1 [week 1]), OLE visits 3 (week 11) and 5 (week 23)
Population: The intent-to-treat (ITT) population (all subjects randomized in the parent study)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 5 | 43 | 17
score on a scale
  visit 1 study 1 | 649.80 (509.54) | 1091.70 (362.11) | 767.47 (227.42)
  OLE visit 0 | 293.60 (243.62) | 376.00 (274.06) | 260.29 (150.02)
  OLE visits 3 | 219.60 (53.07) | 364.53 (272.42) | 113.12 (31.37)
  OLE visits 5 | 179.20 (64.87) | 262.16 (216.67) | 78.94 (20.77)
Statistical Analysis 1: Comparison: Group A vs Group B vs Group C; No sample size calculation was performed. Maximum expected number of participants for OLE was 72 patients randomized to the NOLTREX™ group in the parent study (IA/PAAG-SI/OA/2019). A total of 65 patients entered the OLE. The study did not have a formal hypothesis. The between-group comparison of changes from baseline (OLE visit 0) in the WOMAC-T at visit 5 was conducted using analysis of covariance (ANCOVA) and, as a post hoc test, the Tukey test; Test type: Superiority; p = 0.004, ANCOVA — The threshold for statistical significance was p <0.05; To compare the efficacy of one and two NOLTREX™ courses was used ANCOVA adjusted for the baseline value with fixed factor of "treatment group"; F value = 5.919
Statistical Analysis 2: Comparison: Group A vs Group B; Post-hoc pairwise comparisons were performed using Tukey test; Test type: Superiority; p = 0.783, Tukey's HSD — Difference between Least-square means was tested at a level of p <0.05 via Tukey's multiple comparison test; LS-means difference = -37.64, 95% CI 2-sided [-172.98 to 97.70], Standard Error of Mean 56.34
Statistical Analysis 3: Comparison: Group A vs Group C; Post-hoc pairwise comparisons were performed using Tukey test; Test type: Superiority; p = 0.370, Tukey's HSD; LS-means difference = 81.94, 95% CI 2-sided [-63.28 to 227.16], Standard Error of Mean 60.45
Statistical Analysis 4: Comparison: Group B vs Group C; Post-hoc pairwise comparisons were performed using Tukey test; Test type: Superiority; p = 0.003, Tukey's HSD — Difference between Least-square means was tested at a level of p <0.05 via Tukey's multiple comparison test; LS-means difference = 119.58, 95% CI 2-sided [36.09 to 203.07], Standard Error of Mean 34.76
Statistical Analysis 5: Comparison: Group A vs Group B vs Group C; The between-group comparison of changes from baseline (visit 1 study 1) in the WOMAC-T at visit 5 was conducted using analysis of covariance (ANCOVA) and, as a post hoc test, the Tukey test; Test type: Superiority; p = 0.070, ANCOVA — The threshold for statistical significance was p <0.05; [statistical method as in outcome 1, analysis 1]; F value = 2.78

2. Secondary Outcome: Change in the WOMAC Pain Score (WOMAC-A)
Description: Mean change in WOMAC-A from baseline (visit 1 (week 1) of the parent study AND visit 0 [screening] of OLE) to visit 3 (week 11) and visit 5 (week 23). Patients were asked to complete the questionnaire during the study visits. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a set of standardized questionnaires used by health professionals to evaluate pain, stiffness and physical functioning of the joints in patients with knee and/or hip osteoarthritis. The WOMAC Index Version 3.1 Visual Analog Scale Format (WOMAC VA 3.1) applies a 100 mm VAS. The WOMAC pain scale consists of five items: (1) walking on flat ground; (2) going up or down stairs; (3) at night while in bed; (4) sitting or lying; and (5) standing upright. The scores for the Pain subscale are summed up, with a possible score range of 0-500. Higher scores represent worse pain.
Time Frame: baseline (OLE visit 0 and visit 1 study 1 [week 1]), OLE visits 3 (week 11) and 5 (week 23)
Population: The intent-to-treat (ITT) population (all subjects randomized in the parent study).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 5 | 43 | 17
score on a scale
  visit 1 study 1 | 125.80 (99.55) | 211.02 (77.97) | 158.18 (63.77)
  OLE visit 0 | 60.00 (51.53) | 67.26 (52.72) | 44.24 (28.77)
  OLE visit 3 | 38.00 (18.33) | 65.02 (51.23) | 6.29 (3.89)
  OLE visit 5 | 30.00 (25.67) | 47.98 (44.80) | 3.12 (2.87)

3. Secondary Outcome: Change in the WOMAC Stiffness (WOMAC-B) Score
Description: Mean change in WOMAC-B from baseline (visit 0 [screening] of the OLE and visit 1 [week 1] of the parent study) to visits 3 (week 11) and 5 (week 23). Patients were asked to complete the questionnaire during the study visits. The Western Ontario and McMaster Universities Osteoarthritis Index Version 3.1 Visual Analog Scale Format (WOMAC VA 3.1) applies a 100 mm VAS and consists of three subscales: pain (5 questions), stiffness (2 questions), and physical function (17 questions). The scores for each subscale are summed up, with a possible score range of 0-200 for Stiffness, and 0-1700 for Physical Function. Higher scores represent worse stiffness and functional limitations. The higher the score, the poorer the function. Therefore, an improvement was achieved by reducing the overall score.
Time Frame: baseline (OLE visit 0 and parent study visit 1 [week 1]), visits 3 (week 11) and 5 (week 23)
Population: The intent-to-treat (ITT) population (all subjects randomized in the parent study).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 5 | 43 | 17
score on a scale
  visit 1 study 1 | 78.60 (69.50) | 95.23 (43.13) | 69.94 (26.93)
  OLE visit 0 | 26.00 (30.29) | 30.16 (29.21) | 26.29 (18.11)
  OLE visit 3 | 15.80 (6.83) | 28.05 (29.85) | 21.24 (6.71)
  OLE visit 5 | 12.20 (7.60) | 20.63 (25.03) | 12.12 (4.41)

4. Secondary Outcome: Change in the WOMAC Physical Function (WOMAC-C) Score
Description: Mean change in WOMAC-C from baseline (visit 0 [screening] of the OLE and visit 1 [week 1] of the parent study) to visits 3 (week 11) and 5 (week 23). Patients were asked to complete the questionnaire during the study visits. The Western Ontario and McMaster Universities Osteoarthritis Index Version 3.1 Visual Analog Scale Format (WOMAC VA 3.1) applies a 100 mm VAS and consists of three subscales: pain (5 questions), stiffness (2 questions), and physical function (17 questions). The scores for each subscale are summed up, with a possible score range of 0-200 for Stiffness, and 0-1700 for Physical Function. Higher scores represent worse stiffness and functional limitations. The higher the score, the poorer the function. Therefore, an improvement was achieved by reducing the overall score.
Time Frame: baseline (OLE visit 0 and parent study visit 1 [week 1]), visits 3 (week 11) and 5 (week 23)
Population: The intent-to-treat (ITT) population (all subjects randomized in the parent study)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 5 | 43 | 17
score on a scale
  visit 1 study 1 | 445.40 (364.01) | 785.44 (280.73) | 539.35 (170.29)
  OLE visit 0 | 207.60 (165.18) | 278.58 (200.64) | 189.76 (109.22)
  OLE visit 3 | 165.80 (32.77) | 271.47 (200.43) | 85.59 (24.11)
  OLE visit 5 | 137.00 (37.14) | 193.56 (154.29) | 63.71 (16.15)

5. Secondary Outcome: Change in the 100-mm VAS Pain Score Visual Analogue Scale (100 mm VAS)
Description: Mean change in the VAS pain score from baseline (visit 0 [screening] of the OLE and visit 1 [week 1] of the parent study to visit 2 (week 1), visit 3 (week 11) and visit 5 (week 23). The 0 to 100 mm visual analogue scale (VAS) was used for measuring pain intensity. VAS ratings between 0 and 4 mm were interpreted as no pain, 5 to 44 mm, mild pain; 45 to 74 mm, moderate pain; and 75 to 100 mm, severe pain. The pain VAS was self-completed by the patients.
Time Frame: baseline (OLE visit 0 and study 1 visit 1 [week 1]), OLE visits 3 (week 11) and 5 (week 23)
Population: The intent-to-treat (ITT) population (all subjects randomized in the parent study)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Group A: Group A consisted of 5 patients who received 2 NOLTREX™ courses in the parent study (IA/PAAG-SI/OA/2019) and at Visits 1/2 of OLE (IA/PAAG-SI/OA/2020).
- Group B: Group B comprised 43 patients who received 2 NOLTREX™ courses in the parent study (IA/PAAG-SI/OA/2019) and at Visits 3/4 of OLE.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 5 | 43 | 17
score on a scale
  study 1 visit 1 | 47.20 (19.25) | 58.63 (11.36) | 64.35 (10.86)
  visit 0 | 30.80 (16.33) | 17.33 (10.18) | 9.47 (5.51)
  visit 3 | 11.20 (6.53) | 29.07 (15.29) | 21.53 (6.32)
  visit 5 | 6.20 (5.59) | 16.56 (12.32) | 4.88 (3.14)
Statistical Analysis 1: Comparison: Group A vs Group B vs Group C; BASELINE (study 1 visit 1) To determine a statistically significant difference between 3 groups the one-way ANOVA (for normally distributed data; aov) or the Kruskal-Wallis test (for non-normally distributed data; kw) was used. The Shapiro-Wilk test was employed to assess the normality of the data distribution; Test type: Superiority; p = 0.030, Kruskal-Wallis — The threshold for statistical significance was p <0.05
Statistical Analysis 2: Comparison: Group A vs Group B vs Group C; BASELINE (OLE visit 0) To determine a statistically significant difference between 3 groups the one-way ANOVA (for normally distributed data; aov) or the Kruskal-Wallis test (for non-normally distributed data; kw) was used. The Shapiro-Wilk test was employed to assess the normality of the data distribution; Test type: Superiority; p = 0.002, Kruskal-Wallis — The threshold for statistical significance was p <0.05
Statistical Analysis 3: Comparison: Group A vs Group B vs Group C; visit 3 To determine a statistically significant difference between 3 groups the one-way ANOVA (for normally distributed data; aov) or the Kruskal-Wallis test (for non-normally distributed data; kw) was used. The Shapiro-Wilk test was employed to assess the normality of the data distribution; Test type: Superiority; p = 0.007, ANOVA — The threshold for statistical significance was p <0.05
Statistical Analysis 4: Comparison: Group A vs Group B vs Group C; visit 5 To determine a statistically significant difference between 3 groups the one-way ANOVA (for normally distributed data; aov) or the Kruskal-Wallis test (for non-normally distributed data; kw) was used. The Shapiro-Wilk test was employed to assess the normality of the data distribution; Test type: Superiority; p < 0.001, Kruskal-Wallis — The threshold for statistical significance was p <0.05

6. Secondary Outcome: Patient's Assessment of the Treatment Efficacy
Description: Patient satisfaction with treatment was measured by a 6-point Likert scale (evident aggravation, aggravation, without changes, weak improvement, improvement, significant improvement) at the study visits 3 (week 11) and 5 (week 23).
Time Frame: visits 3 (week 13) and 5 (week 25)
Population: The intent-to-treat (ITT) population (all subjects randomized in the parent study)
Measure: Count of Participants; unit: Participants
Groups:
- Group A: Group A consisted of 5 patients who received 2 NOLTREX™ courses in the parent study IA/PAAG-SI/OA/2019 and at Visits 1/2 of OLE.
- Group B: Group B comprised 43 patients who received 2 NOLTREX™ courses in the parent study and at Visits 3/4 of OLE.
- Group C: Group C consisted of 17 patients who had received 1 NOLTREX™ course in the parent study.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 5 | 43 | 17
Participants
  Visit 3: evident aggravation | 0 | 0 | 0
  Visit 3: aggravation | 0 | 0 | 0
  Visit 3: without changes | 0 | 2 | 5
  Visit 3: weak improvement | 0 | 15 | 8
  Visit 3: improvement | 2 | 23 | 4
  Visit 3: significant improvement | 3 | 3 | 0
  Visit 5: evident aggravation | 0 | 0 | 0
  Visit 5: aggravation | 0 | 0 | 0
  Visit 5: without changes | 0 | 0 | 0
  Visit 5: weak improvement | 0 | 12 | 1
  Visit 5: improvement | 1 | 25 | 16
  Visit 5: significant improvement | 4 | 6 | 0
Statistical Analysis 1: Comparison: Group A vs Group B vs Group C; Fisher's exact test was used to determine whether there is a significant difference between 3 groups. visit 3; Test type: Superiority; p < 0.001, Fisher Exact — The threshold for statistical significance was p <0.05
Statistical Analysis 2: Comparison: Group A vs Group B vs Group C; visit 5 Fisher's exact test was used to determine whether there is a significant difference between 3 groups; Test type: Superiority; p < 0.001, Fisher Exact

7. Secondary Outcome: Investigator's Assessment of the Treatment Efficacy
Description: Investigator satisfaction with treatment was measured by a 6-point Likert scale (evident aggravation, aggravation, without changes, weak improvement, improvement, significant improvement) at the study visits 3 (week 11) and 5 (week 23).
Time Frame: visits 3 (week 13) and 5 (week 25)
Population: The intent-to-treat (ITT) population (all subjects randomized in the parent study).
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 5 | 43 | 17
Participants
  Visit 3: evident aggravation | 0 | 0 | 0
  Visit 3: aggravation | 0 | 0 | 0
  Visit 3: without changes | 0 | 3 | 5
  Visit 3: weak improvement | 1 | 14 | 8
  Visit 3: improvement | 2 | 23 | 4
  Visit 3: significant improvement | 2 | 3 | 0
  Visit 5: evident aggravation | 0 | 0 | 0
  Visit 5: aggravation | 0 | 0 | 0
  Visit 5: without changes | 0 | 1 | 0
  Visit 5: weak improvement | 1 | 11 | 1
  Visit 5: improvement | 0 | 25 | 16
  Visit 5: significant improvement | 4 | 6 | 0
Statistical Analysis 1: Comparison: Group A vs Group B vs Group C; visit 3 Fisher's exact test was used to determine whether there was a significant difference between 3 groups; Test type: Superiority; p = 0.018, Fisher Exact — The threshold for statistical significance was p <0.05
Statistical Analysis 2: Comparison: Group A vs Group B vs Group C; visit 5 Fisher's exact test was used to determine whether there was a significant difference between 3 groups; Test type: Superiority; p < 0.001, Fisher Exact — The threshold for statistical significance was p <0.05

8. Secondary Outcome: Total Number of Paracetamol Tablets Taken
Description: A patient diary was used to capture data about the number of paracetamol 500 mg tablets taken.
Time Frame: visits 3 (week 13) and 5 (week 25)
Population: The intent-to-treat (ITT) population (all subjects randomized in the parent study). The mean number of tablets was calculated taking into account only patients who had received paracetamol.
Measure: Number; unit: paracetamol tablets
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 5 | 43 | 17
paracetamol tablets
  visit 3 | 0 | 0 | 0
  visit 5 | 0 | 0 | 0

9. Secondary Outcome: Total Number of NSAID Tablets Taken
Description: A patient diary was used to capture data about the number of NSAID tablets taken. In case of paracetamol ineffectiveness and pain persistence patient was allowed to take protocol-permitted NSAID at certain doses.
Time Frame: visits 3 (week 11) and 5 (week 23)
Population: The intent-to-treat (ITT) population (all subjects randomized in the parent study)
Measure: Number; unit: NSAID tablets
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 5 | 43 | 17
NSAID tablets
  visit 3 | 0 | 0 | 0
  visit 5 | 0 | 0 | 0

10. Secondary Outcome: The JSN in the Target Knee
Description: Joint space narrowing (JSN) was scored by comparison of subsequent radiographs taken over time. An increase in the radiographic knee JSN is associated with osteoarthritis progression.
Time Frame: baseline (visit 1 of the parent study IA/PAAG-SI/OA/2019), visit 5 (week 23) of OLE
Population: The intent-to-treat (ITT) population (all subjects randomized in the parent study).
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 5 | 43 | 17
millimeters | -0.02 (0.05) | -0.00 (0.19) | 0.02 (0.08)
Statistical Analysis 1: Comparison: Group A vs Group B vs Group C; To determine a statistically significant difference between 3 groups the one-way ANOVA (for normally distributed data; aov) or the Kruskal-Wallis test (for non-normally distributed data; kw) was used. The Shapiro-Wilk test was employed to assess the normality of the data distribution; Test type: Superiority; p = 0.010, Kruskal-Wallis — The threshold for statistical significance was p <0.05

ADVERSE EVENTS:
Time Frame: 6 months from visit 0 to visit 5.
Description: Adverse events are counted in the safety population. The safety population completely overlapped with the ITT population.
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/43 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/43 | 0/17
Other Adverse Events (participants affected / at risk) | 1/5 | 0/43 | 0/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=5) | Group B (N=43) | Group C (N=17)
Suspected coronavirus disease 2019 (COVID-19) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Suspected coronavirus disease 2019 (COVID-19) was considered as apparently not related to the assigned treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT06429319/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT06429319/SAP_001.pdf